CLINICAL TRIAL: NCT01773915
Title: New Proteins in Body Fluids as Potential Biomarker for Alzheimer's Disease: a Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jos Tournoy, MD PhD, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: s54591
Record Dates: First submitted 2012-12-26; First posted 2013-01-23 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Alzheimer Disease, Late Onset
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, blood and saliva in Biobank
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AD patients: Subject fulfilling the McKhann criteria for clinical probable AD
- Healthy elder persons: Healthy controls with abscence of any cognitive disorder

SUMMARY:
Alzheimer's disease (AD) is the most common neurodegenerative disorder afflicting the elderly. Currently, some biochemical tests performed on Cerebrospinal Fluid (CSF) samples have demonstrated to discriminate to some extend between AD and non-AD individuals based on the levels of tau, phospho-tau or Aβ42. We aim to investigate newly identified proteins whose levels increase during the Braak Stages of AD that are accessible in other body fluids such as blood, urine or saliva. The detection of these proteins would allow performing simple tests in case its levels were confirmed to be associated with the AD pathology.

DETAILED DESCRIPTION:
We do not desire to provide a more extensive description

ELIGIBILITY:
Inclusion Criteria:

- mild to moderate AD

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Persons with Alzheimer's disease
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Differences in blood, saliva and urine protein levels in patients with Alzheimer's Disease versus healthy controls. | Up to 1 year
  Protein levels will be measured by classical immunoblotting blot analysis and quantified; Classical statistical analyses will be performed in order to detect any significant differences.

CONTACTS AND LOCATIONS:
Overall Officials: Bart De Strooper, Principal Investigator — KU Leuven; Francesc Guix, Principal Investigator — KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

REFERENCES:
- [Background] Gonzales PA, Pisitkun T, Hoffert JD, Tchapyjnikov D, Star RA, Kleta R, Wang NS, Knepper MA. Large-scale proteomics and phosphoproteomics of urinary exosomes. J Am Soc Nephrol. 2009 Feb;20(2):363-79. doi: 10.1681/ASN.2008040406. Epub 2008 Dec 3. PMID 19056867